CLINICAL TRIAL: NCT06394076
Title: A Multicenter, Evaluator-blinded, Randomized, No-treatment Controlled Study to Evaluate the Safety and Effectiveness of MAILI PRECISE With Lidocaine Injectable Gel for Correction of Infraorbital Hollowing in Chinese Population
Brief Title: A Study to Evaluate the Safety and Effectiveness of Injectable Gel for Correction of Infraorbital Hollowing in Chinese Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinclair Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDM6008A-301
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Infraorbital Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cross-linked sodium hyaluronate gel for injection containing lidocaine (Experimental): Cross-linked sodium hyaluronate gel for injection containing lidocaine
  Interventions: Device: Cross-linked sodium hyaluronate gel for injection containing lidocaine
- No treatment control (No Intervention): No treatment control

INTERVENTIONS:
Device: Cross-linked sodium hyaluronate gel for injection containing lidocaine — Cross-linked sodium hyaluronate gel for injection containing lidocaine
  Arms: Cross-linked sodium hyaluronate gel for injection containing lidocaine

SUMMARY:
A Multicenter, Evaluator-blinded, Randomized, No-treatment Controlled Study to Evaluate the Safety and Effectiveness of MAILI PRECISE With Lidocaine Injectable Gel for Correction of Infraorbital Hollowing in Chinese Population

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above (subject to the time of signing the informed consent form) , gender is not limited;
2. According to Allergan Infraorbital Rim Scale (AIHS), the subjects were judged by blinded evaluator as having "moderate" or "severe" infraorbital rim hallowing (grade 2-3) in each eye, and both eyes must meet the requirements but do not need to have the same score;
3. The injection investigator believes that the hallowing of the infraorbital rim area of the subject can be corrected to grade 0 or grade 1;
4. Able and willing to follow the investigator's guidance, following the treatment restrictions in this protocol, and completing all the visits of this trial as required ;
5. Able to complete the self-assessment of effectiveness without the use of glasses (contact lenses are accepted if the subject wear contact lenses for all the follow-up visits);
6. Volunteer to participate in this clinical trial and sign the Informed Consent Form.

Exclusion Criteria:

1. Atrophy in the infraorbital area;
2. Previous trauma to the infraorbital area, or residual defects, deformities, or scarring in the periorbital or cheek area before screening;
3. The investigator considers that there is a large lower eyelid fat pad that will affect the treatment outcome;
4. The front most part of the eyeball protrudes forward more than the front most part of the cheek;
5. Hyperpigmentation in the infraorbital area (excluding dark circles which are not caused by hyperpigmentation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
At 3 months after the last treatment in the experimental group, and 3 months after the randomization of the control group, blinded evaluators will use AIHS to evaluate the improvement rate of the infraorbital hallowing. | 3 month

SECONDARY OUTCOMES:
At one month after the last injection in the experimental group, and at one month after randomization in the control group, the Allergan Infraorbital Hollowing Scale (AIHS) rating will be evaluated by a blinded investigator | 1 month
At 1 month and 3 months after the last treatment in the experimental group, and at 1 month and 3 months after randomization in the control group, the injection investigator will use AIHS to evaluate the improvement rate of the infraorbital hallowing | 1 month and 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Hongsen Bi, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China